CLINICAL TRIAL: NCT02356900
Title: Effects of High Intensity Interval Training in a Hyperoxic-hyperbaric Environment on Exercise Performance at Altitude
Brief Title: Hyperbaric VO2max Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding required to enroll target subject number
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00060147
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Exercise Training
Keywords: interval training; hyperbaric oxygen; VO2 max; altitude; exercise performance; mitochondrial oxidative capacity; mitochondrial biogenesis
MeSH Terms: interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyperoxic, Hyperbaric (Experimental): Hyperoxic hyperbaric interval exercise training Six sessions of 30 min.of High-intensity interval training completed on a 3-times a week basis at 1.4 ATA of oxygen in a hyperbaric chamber.
  Interventions: Procedure: Hyperoxic hyperbaric interval exercise training; Drug: Oxygen
- Normoxic, Normobaric (Sham Comparator): Normoxic, normobaric, interval exercise training Six sessions of 30 min.of High-intensity interval training completed on a 3-times a week basis.
  Interventions: Procedure: Normoxic, normobaric, interval exercise training

INTERVENTIONS:
Procedure: Hyperoxic hyperbaric interval exercise training — Six 30-min high-intensity interval training sessions completed 3-times a week while at 1.4 ATA of oxygen in a hyperbaric chamber.
  Arms: Hyperoxic, Hyperbaric
Procedure: Normoxic, normobaric, interval exercise training — Six 30-min high-intensity interval training sessions completed 3-times a week.
  Arms: Normoxic, Normobaric
Drug: Oxygen — Used in Hyperoxic hyperbaric interval exercise training intervention
  Arms: Hyperoxic, Hyperbaric

SUMMARY:
This study seeks to examine the effectiveness of training while in a hyperoxic-hyperbaric environment for exercise performance at altitude. Subjects will complete a short, high-intensity interval training (HIT) program inside the hyperbaric chamber.Before and after this training phase, all subjects will be tested for maximum aerobic capacity at a simulated high altitude of 15,000ft in a hypobaric chamber, as well as for molecular markers of mitochondrial oxidative capacity in a skeletal muscle biopsy.

A group of individuals of similar characteristics completing this training program in a normoxic-normobaric environment will serve as a control.

ELIGIBILITY:
Inclusion Criteria:

* healthy, recreationally active or sedentary individuals

Exclusion Criteria:

* VO2max < 35 ml/kg/min - male 30 ml/kg/min - female
* chronic cardiovascular or pulmonary diseases
* history of pneumothorax
* active smoker
* pregnant women
* non-english speaking
* not in full mental capacity
* blind
* sickle cell trait or disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

REFERENCES:
- [Derived] Alvarez Villela M, Dunworth SA, Kraft BD, Harlan NP, Natoli MJ, Suliman HB, Moon RE. Effects of high-intensity interval training with hyperbaric oxygen. Front Physiol. 2022 Aug 19;13:963799. doi: 10.3389/fphys.2022.963799. eCollection 2022. PMID 36060678

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 25 participants were consented. 21 were randomized and completed the study, 1 was a screen failure, 1 withdrew after the initial biopsy and rash from bandage adhesive, 1 was withdrawn due to schedule noncompliance, and one was withdrawn after a syncopal episode during the initial biopsy.
Period: Overall Study
Arm/Group | Hyperoxic, Hyperbaric | Normoxic, Normobaric
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyperoxic, Hyperbaric | Normoxic, Normobaric | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (4.5) | 25.9 (4.8) | 25.4 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 8 | 9 | 17
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximum Aerobic Capacity (VO2max) From Baseline to Post-training (< 72 Hours )
Description: Graded exercise test to exhaustion at simulated 15000 ft altitude
Time Frame: Baseline and <72 hrs Post-training
Population: Three participants in the Hyperoxic, Hyperbaric group and one participant in the Normoxic, Normobaric group were not included in the analysis due to experimental errors.
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Hyperoxic, Hyperbaric | Normoxic, Normobaric
Number analyzed (Participants) | 8 | 9
mL/kg/min | 3.8 (5.0) | 4.2 (4.9)

2. Primary Outcome: Change in Ventilatory Threshold (VT) From Baseline to Post-training (<72 Hours)
Description: Graded exercise test to exhaustion at simulated 15000 ft altitude
Time Frame: Baseline and <72 hrs Post-training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Hyperoxic, Hyperbaric | Normoxic, Normobaric
Number analyzed (Participants) | 8 | 9
mL/kg/min | 3.2 (4.9) | 2.3 (3.4)

3. Primary Outcome: Mitochondrial Mass Change
Description: Immunofluorescence microscopy using citrate synthase staining
Time Frame: Baseline/24 hrs Post-training
Population: Muscle Biopsy samples were not analyzed due to funding issues.
Arm/Group | Hyperoxic, Hyperbaric | Normoxic, Normobaric
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Tfam Muscle Protein Content Change
Description: Western analysis
Time Frame: Baseline/24 hrs Post-training
Population: Muscle Biopsy samples were not analyzed due to funding issues.
Arm/Group | Hyperoxic, Hyperbaric | Normoxic, Normobaric
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Pgc-1a Coactivator Muscle Protein Content Change
Description: Western analysis
Time Frame: Baseline/24 hrs Post-training
Population: Muscle Biopsy samples were not analyzed due to funding issues.
Arm/Group | Hyperoxic, Hyperbaric | Normoxic, Normobaric
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: COX-I Gene Expression Change
Description: Real-time PCR
Time Frame: Baseline/24 hrs Post-training
Population: Muscle Biopsy samples were not analyzed due to funding issues.
Arm/Group | Hyperoxic, Hyperbaric | Normoxic, Normobaric
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Muscle Phenotype Change
Description: Immunofluorescence microscopy using citrate synthase staining
Time Frame: Baseline/24 hrs Post-training
Population: Muscle Biopsy samples were not analyzed due to funding issues.
Arm/Group | Hyperoxic, Hyperbaric | Normoxic, Normobaric
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Hyperoxic, Hyperbaric | Normoxic, Normobaric
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hyperoxic, Hyperbaric (N=11) | Normoxic, Normobaric (N=10)
Dizziness (General disorders) | 0 (0) | 1 (1) — Dizziness resulting from hypoxemia due to exposure to high altitude, 15,000'.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No